CLINICAL TRIAL: NCT00605306
Title: A Randomized, Double-blind, Placebo-controlled, Parallel Group Study to Investigate the Safety and Tolerability of 14-days Treatment With an Inhaled Dose of QMF149 (500/800) in Mild to Moderate Asthmatic Patients
Brief Title: Safety and Tolerability of Indacaterol Maleate/Mometasone Furoate Delivered Via the Twisthaler® Device After 14 Days Treatment in Patients With Mild to Moderate Asthma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CQMF149A2203
Record Dates: First submitted 2008-01-18; First posted 2008-01-31 (Estimated); Results first posted 2013-04-22 (Estimated); Last update posted 2013-04-22 (Estimated); Status verified 2013-03

CONDITIONS: Asthma
Keywords: Asthma; spirometry; lung function; serum cortisol; serum potassium; plasma glucose
MeSH Terms: conditions — Asthma | interventions — Mometasone Furoate; QMF149

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- indacaterol maleate/mometasone furoate (Experimental): Participants received 2 inhalations of indacaterol maleate / mometasone furoate 250/400 μg once daily in the evening (full dose 500/800 μg) delivered via the Twisthaler device for 14 days.
  Interventions: Drug: indacaterol maleate / mometasone furoate
- Placebo (Placebo Comparator): Participants received 2 inhalations of placebo to indacaterol maleate / mometasone furoate once daily in the evening delivered via the Twisthaler device for 14 days.
  Interventions: Drug: placebo to indacaterol maleate/mometasone furoate

INTERVENTIONS:
Drug: indacaterol maleate / mometasone furoate — Indacaterol maleate / mometasone furoate 250/400 μg, 2 puffs once daily delivered via the Twisthaler device.
  Other Names: QMF149
  Arms: indacaterol maleate/mometasone furoate
Drug: placebo to indacaterol maleate/mometasone furoate — Placebo to indacaterol maleate/mometasone furoate delivered via the Twisthaler device.
  Arms: Placebo

SUMMARY:
This study will investigate the safety and tolerability of indacaterol maleate/mometasone furoate via the Twisthaler device after 14 days treatment in patients with mild to moderate asthma.

ELIGIBILITY:
Inclusion Criteria:

* Male and female adult patients aged 18-65 years (inclusive)
* Patients with mild-moderate asthma
* Forced expiratory volume in one second (FEV1) at Visits 1 and 2 are ≥60% of the predicted normal value for the patient.
* Body mass index (BMI) must be within the range of 18-32 kg/m^2.
* Non-smokers or light smokers (≤10 cigarettes per day), with a smoking history of 10 pack years or less.

Exclusion Criteria:

* Patients who suffer from chronic obstructive pulmonary disease (COPD)
* Patients who have been hospitalized or had emergency treatment for an asthma attack in the 6 months prior to study start
* QTcF interval > 450 msec in men and >470 msec in women
* Pregnant women or nursing mothers
* Females of childbearing potential, regardless of whether or not sexually active, if they are not using a reliable form of contraception (surgical contraception or double barrier methods (to be continued for at least two months following last dose) are acceptable).
* History of immunocompromise, including a positive human immunodeficiency virus (HIV)
* A positive Hepatitis B surface antigen (HBsAg) or Hepatitis C test result.
* History of drug or alcohol abuse within 12 months of dosing

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2008-01; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: NOVARTIS, Principal Investigator — Novartis investigator site
Locations (3):
- France (3):
  - Novartis Investigator Site, Neuil
  - Novartis Investigator Site, Paris
  - Novartis Investigator Site, Poitiers

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Indacaterol Maleate/Mometasone Furoate | Placebo
Started | 14 | 14
Completed | 14 | 13
Not Completed | 0 | 1
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Indacaterol Maleate/Mometasone Furoate | Placebo | Total
Number analyzed (Participants) | 14 | 14 | 28
Age Continuous [Mean (Standard Deviation); unit: years] | 31.0 (7.18) | 33.9 (13.35) | 32.4 (10.62)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 6 | 13
  Male | 7 | 8 | 15

OUTCOME MEASURES:

1. Primary Outcome: Participants With Adverse Events
Description: An adverse event (AE) is the appearance or worsening of any undesirable sign, symptom, or medical condition occurring after starting the study drug even if the event is not considered to be related to study drug. Abnormal laboratory values or test results constitute adverse events only if they induce clinical signs or symptoms, are considered clinically significant, or require intervention.
  A serious adverse event (SAE) is defined as an event which is fatal or life-threatening, results in persistent or significant disability/incapacity, constitutes a congenital anomaly/birth defect, requires inpatient hospitalization or prolongation of existing hospitalization, or is medically significant, i.e., defined as an event that jeopardizes the participant or may require medical or surgical intervention to prevent one of the outcomes listed above.
Time Frame: 15 days
Population: All participants
Measure: Number; unit: participants
Arm/Group | Indacaterol Maleate/Mometasone Furoate | Placebo
Number analyzed (Participants) | 14 | 14
participants
  Any adverse event | 9 | 12
  Serious adverse event | 0 | 0
  AE resulting in discontinuation | 0 | 1

2. Secondary Outcome: Levels of Serum Potassium Over Time
Description: At the specified time-points, blood samples were collected for measurement of serum potassium and the samples analyzed by a central laboratory. The end of study visit was conducted approximately 5-9 days after the last dose.
Time Frame: Baseline; Days 1 and 14 at pre-dose, 0.25, 0.5, 1, 2, 4 hours post-dose; 12 and 24 hours post-dose (Day 2); study completion (5-9 days after last dose, Day 19-23).
Population: All participants
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Indacaterol Maleate/Mometasone Furoate | Placebo
Number analyzed (Participants) | 14 | 14
mmol/L
  Baseline (N=14, 14) | 4.271 (0.2867) | 4.336 (0.3388)
  Day 1, pre-dose (N=14, 14) | 4.264 (0.2240) | 4.279 (0.3446)
  Day 1, 0.25 hours post-dose (N=14, 14) | 4.293 (0.3583) | 4.314 (0.5803)
  Day 1, 0.5 hours post-dose (N=14, 14) | 4.150 (0.2442) | 4.179 (0.3093)
  Day 1, 1 hour post-dose (N=14, 14) | 4.143 (0.2174) | 4.171 (0.2614)
  Day 1, 2 hours post-dose (N=14, 14) | 4.157 (0.2709) | 4.093 (0.2200)
  Day 1, 4 hours post-dose (N=14, 14) | 3.979 (0.2486) | 3.929 (0.2494)
  Day 2, 12 hours post-dose (N=14, 14) | 4.436 (0.2530) | 4.500 (0.2961)
  Day 2, 24 hours post-dose (N=14, 14) | 4.293 (0.2786) | 4.386 (0.4753)
  Day 14, pre-dose (N=14, 14) | 4.150 (0.3205) | 4.136 (0.3079)
  Day 14, 0.25 hours post-dose (N=14, 13) | 4.064 (0.3522) | 4.092 (0.3353)
  Day 14, 0.5 hours post-dose (N=14, 13) | 3.986 (0.3325) | 4.092 (0.3378)
  Day 14, 1 hour post-dose (N=14, 13) | 3.986 (0.3880) | 4.038 (0.4426)
  Day 14, 2 hours post-dose (N=14, 13) | 3.986 (0.2627) | 4.038 (0.3927)
  Day 14, 4 hours post-dose (N=14, 13) | 3.800 (0.3397) | 3.792 (0.2397)
  End of study (N=14, 14) | 4.364 (0.2373) | 4.429 (0.4103)

3. Secondary Outcome: Levels of Plasma Glucose Over Time
Description: At the specified time-points, blood samples were collected for measurement of plasma glucose and the samples analyzed by a central laboratory. The end of study visit was conducted approximately 5-9 days after the last dose.
Time Frame: Baseline; Days 1 and 14 at pre-dose, 0.25, 0.5, 1, 2, 4 hours post-dose; 12 and 24 hours post dose (Day 2); study completion (5-9 days after last dose, Day 19-23).
Population: All participants
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Indacaterol Maleate/Mometasone Furoate | Placebo
Number analyzed (Participants) | 14 | 14
mmol/L
  Baseline (N=14, 14) | 5.079 (0.3239) | 5.157 (0.4415)
  Day 1, pre-dose (N=14, 14) | 5.057 (0.2533) | 5.236 (0.3855)
  Day 1, 0.25 hours post-dose (N=14, 14) | 5.007 (0.2786) | 5.264 (0.4069)
  Day 1, 0.5 hours post-dose (N=14, 14) | 4.950 (0.2279) | 5.207 (0.3385)
  Day 1, 1 hour post-dose (N=14, 14) | 5.036 (0.2620) | 5.193 (0.3316)
  Day 1, 2 hours post-dose (N=14, 14) | 5.057 (0.2377) | 5.179 (0.3142)
  Day 1, 4 hours post-dose (N=14, 14) | 7.064 (1.4532) | 6.793 (1.2344)
  Day 2, 12 hours post-dose (N=14, 14) | 5.221 (0.2326) | 5.286 (0.3009)
  Day 2, 24 hours post-dose (N=14, 14) | 5.293 (0.4463) | 5.321 (0.5767)
  Day 14, pre-dose (N=14, 14) | 5.129 (0.4681) | 5.221 (0.3534)
  Day 14, 0.25 hours post-dose (N=14, 13) | 5.136 (0.4986) | 4.900 (0.4301)
  Day 14, 0.5 hours post-dose (N=14, 13) | 5.157 (0.4767) | 4.946 (0.4409)
  Day 14, 1 hour post-dose (N=14, 13) | 5.136 (0.4448) | 4.962 (0.3841)
  Day 14, 2 hours post-dose (N=14, 13) | 5.093 (0.3269) | 4.908 (0.4173)
  Day 14, 4 hours post-dose (N=14, 13) | 6.929 (1.3176) | 7.408 (1.0649)
  End of study (N=14, 13) | 5.257 (0.2821) | 5.731 (1.0160)

4. Secondary Outcome: Levels of Serum Cortisol Over Time
Description: At the specified time-points, blood samples were collected for measurement of serum cortisol and the samples analyzed by a central laboratory. The end of study visit was conducted approximately 5-9 days after the last dose.
Time Frame: Baseline; Days 1 and 14 at pre-dose, 0.25, 0.5, 1, 2, 4, 11, 12, 13 hours post-dose; 24 hours post dose (Day 2); study completion (5-9 days after last dose, Day 19-23).
Population: All participants
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Indacaterol Maleate/Mometasone Furoate | Placebo
Number analyzed (Participants) | 14 | 14
mmol/L
  Baseline (N=14, 14) | 466.214 (178.2311) | 441.143 (97.5365)
  Day 1, pre-dose (N=14, 14) | 159.643 (100.4533) | 140.714 (47.2024)
  Day 1, 0.25 hours post-dose (N=14, 14) | 153.786 (87.5313) | 151.000 (91.2798)
  Day 1, 0.5 hours post-dose (N=14, 14) | 130.143 (74.2375) | 130.571 (63.6779)
  Day 1, 1 hour post-dose (N=14, 14) | 99.143 (54.5412) | 131.929 (51.4923)
  Day 1, 2 hours post-dose (N=14, 14) | 65.357 (33.1143) | 84.286 (27.1220)
  Day 1, 4 hours post-dose (N=14, 14) | 55.929 (24.6716) | 102.071 (54.8248)
  Day 2, 11 hours post-dose (N=14, 14) | 362.500 (159.3891) | 478.214 (121.2272)
  Day 2, 12 hours post-dose (N=14, 14) | 289.929 (96.3906) | 404.214 (123.4623)
  Day 2, 13 hours post-dose (N=14, 14) | 335.214 (150.7811) | 370.071 (105.2451)
  Day 2, 24 hours post-dose (N=14, 14) | 136.857 (75.4442) | 193.500 (87.5238)
  Day 14, pre-dose (N=14, 14) | 126.071 (65.6546) | 122.857 (71.5379)
  Day 14, 0.25 hours post-dose (N=14, 13) | 111.500 (82.9001) | 127.231 (104.5834)
  Day 14, 0.5 hours post-dose (N=14, 13) | 99.500 (68.5608) | 121.154 (112.2726)
  Day 14, 1 hour post-dose (N=14, 13) | 82.786 (57.7663) | 106.385 (118.7936)
  Day 14, 2 hours post-dose (N=14, 13) | 62.071 (44.5861) | 94.154 (133.8300)
  Day 14, 4 hours post-dose (N=14, 13) | 48.214 (34.5280) | 102.154 (80.7051)
  Day 15, 11 hours post-dose (N=14, 14) | 242.143 (177.3739) | 417.000 (100.8312)
  Day 15, 12 hours post-dose (N=14, 13) | 255.500 (154.1442) | 388.769 (104.6885)
  Day 15, 13 hours post-dose (N=14, 13) | 324.857 (179.8713) | 385.769 (126.2301)
  End of study (N=14, 14) | 495.286 (259.2054) | 417.786 (164.1046)

ADVERSE EVENTS:
Arm/Group | Indacaterol Maleate/Mometasone Furoate | Placebo
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/14
Other Adverse Events (participants affected / at risk) | 9/14 | 12/14
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Indacaterol Maleate/Mometasone Furoate (N=14) | Placebo (N=14)
Blepharitis (Eye disorders) | 0 | 1
Conjunctivitis (Eye disorders) | 0 | 1
Chest discomfort (General disorders) | 0 | 2
Chills (General disorders) | 0 | 1
Bronchitis (Infections and infestations) | 2 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0
Rhinitis (Infections and infestations) | 2 | 2
Tracheitis (Infections and infestations) | 1 | 0
Peak expiratory flow rate decreased (Investigations) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Aphonia (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 5 | 2
Syncope vasovagal (Nervous system disorders) | 0 | 1
Tremor (Nervous system disorders) | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Asthmatic crisis (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 4
Painful respiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.